CLINICAL TRIAL: NCT03051178
Title: Wearable Sensor Driven Closed-loop Deep Brain Stimulation for Essential Tremor
Brief Title: Wearable Sensor for Responsive DBS for ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medtronic (Industry); De Luca Foundation (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201602458 -A; OCR17477 (Other: UF OnCore); 1F31NS115363-01A1 (NIH); UH3NS095553 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-10

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with Essential Tremor (Experimental): This cohort will receive deep brain stimulation (DBS) therapy responsively based on the level of their symptoms as detected by wearable EMG and inertia (acceleration) sensors.
  Interventions: Device: Responsive deep brain stimulation

INTERVENTIONS:
Device: Responsive deep brain stimulation — Responsive deep brain stimulation (R-DBS) therapy will be delivered responsively based on the level of their symptoms as detected by wearable EMG and inertia (acceleration) sensors.

SUMMARY:
The purpose of this study is evaluate the effectiveness and safety of a possible new treatment for Essential Tremor (ET) using external wearable sensors, which have the capability of recording acceleration and Electromyography (EMG). This therapy is called Responsive Deep Brain Stimulation (R-DBS). R-DBS systems will communicate with a computer, and apply stimulation when the computer detects patterns associated with tremor. This detection will suppress pathological activity and improve or alleviate the tremor.

Currently, DBS is approved for the treatment of ET; however, stimulation is delivered continuously even when tremor or other symptoms are absent. Continuous DBS can lead to unwanted side effects such as stuttering and gait\balance problems. On the other hand, R-DBS will turn on only if activity associated with ET from the external sensors is detected.

DETAILED DESCRIPTION:
The overall purpose of this application is to capture pathological activity related to essential tremor using external wearable sensors to responsively initiate or terminate DBS. To this end, the researchers propose to use the Nexus-D system, which requires a firm ware update to an Activa Implantable Neurostimulator (INS), and it will in a smart way turn DBS on/off in patients. The study team will recruit subjects with Activa SC or PC neurostimulator implants during 6 post-operative programming visits. The research group is already familiar with and is in possession of the Nexus-D system, and the investigators have successfully performed responsive DBS in two patients with Tourette syndrome (TS) and in four patients with Parkinson's disease in acute settings. The lab is also equipped with wireless wearable sensor and amplifier systems, such as a 16-unit wireless EMG+ acceleration+inertia Trigno Wireless Bio Acquisition System (Delsys Inc, Natick, MA). The study team aims to combine these signal modalities to capture pathological symptoms and generate commands to initiate or terminate DBS (also record adverse side effects, if any). The project goal is to characterize the clinical efficacy, side effect profile, and battery life of closed-loop DBS in acute settings using wearable sensors in essential tremor patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Patient is over 21 years of age
* Patient has had a significant disabling, medication-refractory upper extremity tremor with no evidence of non-ET central nervous system disease or injury for at least three (3) months prior to implantation of Activa SC, PC, or RC device.
* Patient receives Vim electrode and Activa SC, PC or RC device implants, and recovers fully after surgery.
* Patient is available for study participation after their clinical programming appointments for six months.

Exclusion Criteria:

* Medication related movement disorders.
* Any suspicion of Parkinsonian tremor, including presence of Parkinsonian features such as bradykinesia, rigidity, or postural instability.
* Severe medical co-morbidity including cardiovascular disorder, lung disorder, kidney disease, continuous neurological disease, hematological disease, or frailty that impact tolerability of the surgery as judged by the screening physicians.
* Patient is undergoing a lead revision surgery.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gunduz, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health, Gainesville, Florida
  - Biomedical Sciences Building, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 patients were enrolled into the single arm study. 5 patients withdrew from the study. We are comparing their clinical Tremor Rating Scores (TRS) for three conditions: deep brain stimulation (DBS) OFF, standard (continuous) DBS, and responsive DBS (the trial condition).
Period: Overall Study
Arm/Group | Subjects With Essential Tremor
Started | 17
Implementation of Responsive DBS Based on Wearable Sensors | 12
Completed | 12
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Subjects With Essential Tremor: This cohort will receive deep brain stimulation (DBS) therapy responsively based on the level of their symptoms as detected by wearable EMG and inertia (acceleration) sensors.
  Responsive deep brain stimulation: Responsive deep brain stimulation (R-DBS) therapy will be delivered responsively based on the level of their symptoms as detected by wearable EMG and inertia (acceleration) sensors.
  The clinical tremor rating scale (TRS) with R-DBS will be compare to no DBS and continuous DBS TRS scores.
Arm/Group | Subjects With Essential Tremor
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 74.2 [64 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Clinical Rating Scale for Tremor (CRST)
Description: Responsive deep brain stimulation as an effective alternative to continuous deep brain stimulation. Clinical Tremor Rating Scale (TRS), rated by a blinded neurologist, during responsive brain stimulation will be compared to scores during continuous deep brain stimulation and no stimulation. The minimum and maximum score range for this scale is 0-80, with higher score indicating worse outcome.
Time Frame: 30 minutes during one monthly visit after clinical continuous deep brain stimulation is optimized.
Population: We statistically compared the Tremor Rating Scale (TRS) scores for responsive deep brain stimulation (R-DBS) to standard continuous DBS (cDBS) and to NO DBS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects With Essential Tremor
Number analyzed (Participants) | 12
score on a scale
  DBS Off | 18.39534884 (9.191454455)
  Continuous DBS | 13.97674419 (5.616677429)
  Responsive DBS | 14.58139535 (5.197217929)
Statistical Analysis 1: Comparison: Subjects With Essential Tremor; TRS scores measured across different stimulation conditions were assessed using a mixed model ANOVA with the participant as a random effect. All post-hoc comparisons were Bonferroni corrected; Test type: Superiority; p < 0.01, ANOVA — All post-hoc comparisons were Bonferroni corrected

ADVERSE EVENTS:
Time Frame: Adverse events for R-DBS were observed through study completion: 30 minutes during one monthly visit in addition to a 2 week follow up.
Description: We use the same definition of adverse and serious adverse events as clinicaltrials.gov
Arm/Group | Subjects With Essential Tremor
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/78/NCT03051178/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03051178/ICF_001.pdf